CLINICAL TRIAL: NCT03662464
Title: ESCAPE STUDY : A Specific Tool for Detecting Nursing Home Residents (With or Without Dementia) at Risk of Escaping for the Use of Caregivers: Psychometric Properties and Definition of Risk Levels
Brief Title: ESCAPE Study : Validation of a Specific Tool Scoring Residents at Risk of Escaping/Elopement From Nursing Homes (ESCAPE)
Acronym: ESCAPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-55; IDRCB (Other: 2017-A02827-46)
Record Dates: First submitted 2018-08-31; First posted 2018-09-07 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-01

CONDITIONS: Elopement or Escaping of Nursing Home Resident With or Without Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — develop and validate a specific tool to score the risk of escaping in Nursing Homes residents

SUMMARY:
Residents' escapes occur even if most of the nursing homes (NH) have set up specific devices to prevent from this risk. Therefore, the need to develop and validate a specific tool to assess the risk of escaping was obvious to the working group, aim at emphasizing patient centered-care by the nurses' staff and help to develop personalized devices.

Aim of the study: develop and validate a specific tool to score the risk of escaping in NH residents Study design: Observational prospective multicentered cohort study Nursing homes volunteer to participate Location: Provence Alpes Cotes d'Azur Region ( South East of France) Population: 4050 NH residents. Duration: two years, each resident included is followed up for one year Measures: Nursing homes characteristics, residents characteristics ( social and from medical record); Escape Scale (25 items with a Yes/no answer; filled up during a nurses staff meeting for each resident and every three months; 3 sub scales: resident environmental items, social items, and medical items.

ELIGIBILITY:
Inclusion Criteria:

* Every resident of Nursing home participating to the study
* Living in the NH for three months or more
* With a living prognosis longer than 3 Months

Exclusion Criteria:

* Prognosis less than three months
* Bedridden (not able to move alone from bed to chair)
* Nursing home short stay scheduled < 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Resident of the nursing homes in Provence Alpes Cotes d'Azur Region ( South East of France)
Sampling Method: Probability Sample
Enrollment: 4050 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Escape/elopement occurence | 2 years
  Each Event occurrence is notify by the nurses staff at any time

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — Assitance Publique des Hopitaux de Marseille
Locations (1):
- Direction Recherche clinique et Innovation, Marseille, PACA, France